CLINICAL TRIAL: NCT06177899
Title: A Novel Approach for Horizontal Augmentation With Split Box: A Method That Combines Split Bone Block and Ridge Split Techniques
Brief Title: A Novel Approach for Horizontal Augmentation: A Split Box
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: spltbx
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Alveolar Bone Loss; Alveolar Ridge Augmentation; Augmentation, Alveolar Ridge
Keywords: Alveolar ridge augmentation; Horizontal augmentation; Bone block augmentation
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Split-box group: Before augmentation, according to the 3D topography of the alveolar ridge of the patients, the split-box technique was applied if there was more than 3 mm bone thickness at the top of the crest and the bone thickness did not increase towards the lower border.
  All surgical procedures were performed under local anesthesia. A mid-crestal incision was made along the ridge crest and two vertical incisions were made at the termination of the crestal incision. All osteotomies were made using with piezoelectric surgery. Horizontal and vertical osteotomies were performed 1.5 mm away from adjacent teeth. Lower border osteotomy of the vestibular cortical bone was performed. A chisel osteoma was used to separate completely and mobilize the segmented bone. This separated, corticocancellous block was stabilized on the distance to the native alveolar crest with micro screws. The space between the block and the alveolar crest was filled with allograft. The flaps were closed using 3-0,4-0 vicryl.
  Interventions: Procedure: Splitting of bone and fixation of bone laminae differ between the 3 groups.
- Reverse split-box group: Before augmentation, according to the 3D topography of the alveolar ridge of the patients, the reverse split-box technique was applied if there was more than 3 mm bone thickness at the top of the crest and the bone thickness increase towards the lower border.
  This technique differs from the split-box technique as follows: If the bone thickness of the alveolar crest is thick enough to be split, in addition to the bone thickness increases toward the lower border at the alveolar bone, it involves reversing the separated corticocancellous bone block before fixation.
  Interventions: Procedure: Splitting of bone and fixation of bone laminae differ between the 3 groups.
- Sliding split-box group: Before augmentation, according to the 3D topography of the alveolar ridge of the patients, the sliding split-box technique was applied if there was less than 3 mm bone thickness at the top of the crest and the bone thickness increase towards the lower border.
  This technique differs from the split-box technique as follows: If the bone thickness of the alveolar crest is not thick enough to split at the alveolar crest (<3 mm), but the bone thickness increases toward the lower border of the alveolar bone, horizontal osteotomy is performed at the level where the bone thickness reaches at least 3 mm. Separated corticocancellous bone block is slid toward the coronal of alveolar crest and fixed in line with the native alveolar bone.
  Interventions: Procedure: Splitting of bone and fixation of bone laminae differ between the 3 groups.

INTERVENTIONS:
Procedure: Splitting of bone and fixation of bone laminae differ between the 3 groups. — In split-box technique, all osteotomies were made using with piezoelectric surgery. Horizontal and vertical osteotomies were performed 1.5 mm away from adjacent teeth. Lower border osteotomy of the vestibular cortical bone was performed. A chisel osteoma was used to separate completely and mobilize the segmented bone. This separated, corticocancellous block was stabilized on the distance to the native alveolar crest with micro screws. The space between the block and the alveolar crest was filled with allograft. In reverse split box technique, differs from the split-box technique as follows: it involves reversing the separated corticocancellous bone block before fixation. In sliding split box technique, differs from the split-box technique as follows: horizontal osteotomy is performed at the level where the bone thickness reaches at least 3 mm. Separated corticocancellous bone block is slid toward the coronal of alveolar crest and fixed in line with the native alveolar bone.

SUMMARY:
The goal of this clinical study is to investigate the effectiveness of the split-box technique in systemically healthy, non-smoking, over 18 years of age, participants with narrow crests (<5mm bone width) and adequate bone height (>12mm). The main questions it aims to answer are:

* The primary objective of the present study is to investigate the effectiveness of the split-box technique by evaluating the change in width and height of the alveolar bone.
* The secondary objective is to evaluate the superiority of the split-box technique and its modifications in terms of the amount of bone gain.

According to the 3D topography of the alveolar ridge of the patients before augmentation, split box or one of its modifications, reverse split box or sliding split box techniques were selected and applied. (split box was applied if the bone thickness was more than 3 mm at the top of the crest and did not increase towards the lower border at the alveolar bone, reverse split box technique was applied if the bone thickness was more than 3 mm at the top of the crest and increased towards the lower border at the alveolar bone, sliding split box was applied if the bone thickness was less than 3 mm at the top of the crest but the bone thickness increases towards the lower border at the alveolar bone.)

ELIGIBILITY:
Inclusion Criteria:

* To be older than 18 years of age
* To be systemically healthy
* To be non-smokers
* Having narrow crests (<5 mm bone width)
* Having adequate bone height (>12 mm)
* Having cone-beam computed tomography scans before surgery and five months after augmentation

Exclusion Criteria:

* Having bone diseases,
* A history of neck or head radiotherapy
* Receiving steroids, bisphosphonates or chemotherapeutic drugs
* Being pregnancy
* Having narrow bone thickness in the crest (<3 mm), those in whom this thickness did not increase toward the lower border of the alveolar bone
* Patients with a history of infection or exposure after augmentation

Ages: 22 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients whose thickness at the top of the alveolar crest is insufficient for implant placement and who require bone augmentation.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Horizontal changes in the alveolar bone | 5 months
  To determine the horizontal changes in the alveolar bone, thickness was measured at two different levels. The measurements were titled as follows: crestal width (CW) and screw level width (SLW).
  To measure CW, measurements were made horizontally at the highest point of the crest in pre- and post-operative tomography. To measure SLW, in the post-operative tomography, the bone thickness at the screw level was measured horizontally and recorded. In addition, the distance between the anatomical landmark (mandibular basis, mandibular foramen, lower border of nasal or sinus cavity) and the screw level was also measured and recorded. The main goal of this measurement was to provide a reference for SLW measurement on preoperative cone-beam computed tomography (CBCT), since there were no screws. After the measurements in the postoperative CBCT were made, SLW was also made in the preoperative imaging.
Vertical changes in the alveolar bone | 5 months
  To determine whether there was vertical bone loss during horizontal augmentation, the height of the alveolar ridge (ARH) was measured. To measure ARH, a line was created between the anatomical landmark and the highest point of the crest, and the length of this line was measured in the pre- and post-operative tomography.

SECONDARY OUTCOMES:
Difference in bone thickness gain at the top of the crest (CW) between the 3 groups | 5 months
  In order to determine the difference between the 3 groups in terms of CW, the difference between the pre- and post-operative values of the 3 groups was determined. These values were compared between the 3 groups.
Difference in bone thickness gain at the top of the screw level (SLW) between the 3 groups | 5 months
  In order to determine the difference between the 3 groups in terms of SLW, the difference between the pre- and post-operative values of the 3 groups was determined. These values were compared between the 3 groups.
Difference in bone loss at alveolar ridge height (ARH) between 3 groups | 5 months
  In order to determine the difference between the 3 groups in terms of ARH, the difference between the pre- and post-operative values of the 3 groups was determined. These values were compared between the 3 groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided